CLINICAL TRIAL: NCT06783582
Title: Effect of Motivational Interviewing Based on Pender's Health Promotion Model on Patient-Reported Outcomes in Patients With COPD
Brief Title: Effectiveness of Motivational Interviewing in Patients With COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zeynep Yildirim (Other)
Responsible Party: Sponsor-Investigator, Zeynep Yildirim, Research Assistant, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Thesis
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: COPD; Nurse-Patient Relations
Keywords: Patient-reported Outcomes; Nurse; COPD; Motivational Interviewing; Pender's Health Promotion Model
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interviewing (Experimental): The intervention group will given 30-45 minutes of motivational interviewing.
  Interventions: Other: Motivational interviewing based on Pender's health promotion model
- Control Group (No Intervention): Routine nursing care was given to COPD patients in this group without any interview.

INTERVENTIONS:
Other: Motivational interviewing based on Pender's health promotion model — In addition to routine nursing care, patients will be given a motivational interview intervention based on Pender's health promotion model. This intervention will be carried out in a total of 6 sessions, three face-to-face sessions and three online sessions planned individually for each patient. The interviews will last approximately 30-45 minutes. The first motivational interview will be held on the 1st day of the patient's admission to the clinic, the second motivational interview on the 4th day, and the third motivational interview on the 7th day. The face-to-face sessions will be conducted by the researcher in the hospital's education room and contact information will be obtained from the patients. The following three interviews will be held online with the patients once a week via the WhatsApp application. The patient will be contacted at least two days before the interviews, an appointment will be made, and the interview day and time will be determined.
  Arms: Motivational Interviewing

SUMMARY:
To determine the effect of motivational interviewing based on Pender's health promotion model on patient-reported outcomes in patients with COPD.

DETAILED DESCRIPTION:
Nursing, which arises from human needs, evaluates the individual, family, and society with a holistic perspective to protect, maintain, and improve the health of healthy/sick individuals, families, and communities, and provides the necessary health services. The primary duty of nurses is to provide care for individuals and improve their quality of life. In this regard, nurses fulfill their duties by using their roles such as counselor, educator, decision-maker, manager, researcher, and caregiver. Nurses have significant responsibilities in the care of chronic diseases that require lifelong care and follow-up.

One of the major chronic diseases requiring lifelong care is Chronic Obstructive Pulmonary Disease (COPD). COPD is a progressive, irreversible disease characterized by airflow obstruction, accompanied by various symptoms, and is a serious health problem with high mortality and morbidity, commonly encountered worldwide. Approximately 3.2 million people die annually from COPD globally, and it is projected that this disease will be the third leading cause of death worldwide by 2030. COPD patients experience many physical and psychological issues that severely affect their quality of life, such as fear of death, anxiety, cough, dyspnea, fatigue, and loss of appetite . COPD patients are frequently hospitalized, face difficulties in performing daily activities, encounter social and economic losses, and experience a significant decline in quality of life due to the side effects of medications.

Among the long-term management goals of disease control are the reduction of current symptoms and future risks. These goals require patients to exhibit healthy behaviors. However, the literature reports that COPD patients have low levels of self-care, poor adherence to medications, and a lack of awareness regarding preventable and behavioral causal factors. COPD patients need strategies that will engage them in the treatment process, motivate them toward healthy habits, and help internalize healthy behaviors. Compared to other strategies, motivational interviewing (MI) embodies most of these qualities. MI is defined as "collaborative, person-centered form of guiding and counseling to elicit and strengthen motivation for change". The MI technique is a distinctive and superior approach to other interview methods due to its effectiveness in helping individuals make behavioral changes, its empathetic and collaborative approach, its ability to increase intrinsic motivation, and its strategies for dealing with resistance. MI aims to promote change by increasing the patients intrinsic motivation, making it especially effective for patients with more specific change goals.

The use of nursing models in the care of COPD patients has been associated with better patient outcomes, higher nurse satisfaction, and lower healthcare costs. Pender's Health Promotion Model (HPM) provides nurses with a comprehensive framework for conducting effective care and assessing individuals perceptions of health behaviors. The model assumes that individuals have a holistic structure in their physical environment and interpersonal relationships and play an active role in maintaining and promoting their health. The goal of the model is to explain the components of behaviors necessary for a healthy lifestyle, evaluate individuals experiences, analyze factors that may affect their perceptions of health behavior, and guide care providers in planning healthy lifestyle goals. In light of this information, it is recognized that MI and HPM share common goals and possess complementary dynamics. Addressing lifestyle changes with Pender's model and integrating MI for health promotion has been reported to be more effective in managing COPD patients symptoms. Dişsiz and Çalışkan also suggest that nurses can use HPM and MI, which are thought to complement each other, while helping patients acquire healthy lifestyle behaviors.

Patient-reported outcomes are necessary to assess the symptoms, the impact of symptoms on their lives, and their response to treatment. Patient-reported outcomes provide direct reports of patients perceived health statuses. While the primary role of nurses is caregiving, they should also engage in roles such as educator, therapist, counselor, and researcher to implement interventions that improve the care of COPD patients. Nurses should support individuals to use their potential strengths and help them adopt health behaviors through health promotion programs. MI and the Health Promotion Model have been shown to be effective strategies and models in facilitating health behavior change. Based on this information, this research was conducted to determine the effect of motivational interviewing based on Pender's Health Promotion Model on patient-reported outcomes in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age,
* Volunteering to participate in the study,
* Being literate,
* Having GOLD Stage II and III COPD,
* Receiving COPD treatment for more than 6 months,
* Having a smartphone for online interviews,
* Not having sensory loss related to hearing and vision,
* Not having a history of psychiatric diagnosis,
* Being suitable for applying cognitive level scales.

Exclusion Criteria:

* Having GOLD Stage I and IV COPD,
* Having serious pulmonary and malignant disease,
* Not being able to communicate in Turkish,
* Being in an exacerbation period,
* Having a history of psychiatric diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-29 (Actual); Primary Completion 2025-02-24 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Adapted Patient Reported Outcome Scale for Chronic Obstructive Pulmonary Disease | Up to 4 weeks
  The Turkish validity and reliability study of the scale developed by Liu et al. in 2020 was conducted by Sazak and Orgun in 2023. The scale consists of 27 items in three dimensions. The dimensions are physical domain, environmental domain and psychological domain. The scale is a 5-point Likert type (Never 0, Almost never 1, A few times 2, Many times 3, Almost always 4). Item 13 should be reverse scored. Cronbach's Alpha reliability coefficient of the scale was determined as 0.954 for the overall scale, 0.945 for the physical domain sub-dimension, 0.862 for the psychological domain sub-dimension and 0.828 for the environmental sub-dimension.
Modified Medical Research Council (mMRC) Dyspnea Scale | Up to 4 weeks
  The dyspnea scale, developed by Fletcher in 1952, was used to compare the dyspnea levels of individuals with lung disease and those without during activity. Later, the scale was developed by the British Medical Research Council (MRC) to evaluate the course of diseases. The scale, which is based on various physical activities to determine dyspnea, consists of 5 items and is scored between 0 and 4 points. The best point in terms of dyspnea on the scale is 0, while the worst is defined as 4 points.
COPD Assessment Test (CAT) | Up to 4 weeks
  Developed by Jones et al. in 2009, the scale was validated in Turkish by Yorgancıoğlu et al. in 2012. CAT determines disease severity by evaluating symptoms such as cough, phlegm, shortness of breath, fatigue, and leaving home. The scores of the questions in the test range from "0-40". CAT assessment test score; 0-10 is considered "low impact", 11-20 is considered "moderate impact", 21-30 is considered "high impact", and 31-40 is considered "very high impact".

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)